CLINICAL TRIAL: NCT06586138
Title: Study of Psychological, Sociological and Professional Factors Associated With Maintenance of Wakefulness Tests Results
Brief Title: Study of Psychological, Sociological and Professional Factors Associated With Maintenance of Wakefulness Test
Acronym: STAYAWAKE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0658
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: Narcolepsy; Obstructive Sleep Apnea (OSA)
Keywords: Obstructive Sleep Apnea; Maintenance of Wakefulness Test (MVT); Anxiety; Alertness; Sleepiness; Narcolepsy
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive; Anxiety Disorders; Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance of Wakefulness Test: Consecutive patients referred for Maintenance of Wakefulness test at the center for Sleep Medicine in Lyon University hospital (HCL - Croix Rousse Hospital)
  Interventions: Other: STAI (State-Trait Anxiety Inventory) Scale : Psychological inventory of 20 self-report items on a 4-point scale

INTERVENTIONS:
Other: STAI (State-Trait Anxiety Inventory) Scale : Psychological inventory of 20 self-report items on a 4-point scale — Patient completed STAI Scale in the 24 hours before Maintenance of Wakefulness Test during the hospitalization

SUMMARY:
The predictors of objective impaired alertness assessed by Maintenance of Wakefulness Tests (MWT) are poorly understood. Identifying such predictors are essential from a clinical point of view and from a pathophysiological perspective, to better understand the determinants of residual Excessive Daytime Sleepiness (EDS) and the complex link between subjective and objective impairments.

Also, the objective of this study is to describe psychological but also sociological and professional factors associated with Maintenance of Wakefulness Tests results.

ELIGIBILITY:
Inclusion Criteria:

* Adult (i.e. age ≥ 18 y.o)
* referred for Maintenance of Wakefulness test at Lyon University hospital (HCL - Croix Rousse Hospital)

Exclusion Criteria:

* do not consent
* unable to answer the questionary
* cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for Maintenance of Wakefulness test at the center for Sleep Medicine in Lyon University hospital (HCL - Croix Rousse)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) score | baseline
  STAI ((State-Trait Anxiety Inventory) scale is a psychological inventory of 20 self-report items on a 4-point scale. Minimum Score is 20 and maximum score is 80.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine du Sommeil - Hopital Croix Rousse, Lyon, France